CLINICAL TRIAL: NCT04862338
Title: Pharmacodynamics and Tolerance Study of Nicotinamide Mononucleotide (NMN) Supplementation at 400 mg/Day
Brief Title: Pharmacodynamics and Tolerance of Nicotinamide Mononucleotide (NMN, 400mg/Day) in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seneque SA (Industry)
Collaborators: CEN Biotech (Industry); LGD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C1677
Record Dates: First submitted 2021-04-21; First posted 2021-04-28 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
Keywords: tolerance; Pharmacodynamics
MeSH Terms: interventions — Nicotinamide Mononucleotide

STUDY DESIGN:
Intervention Model Description: Exploratory interventional repeated-dose study, open-label, single-arm, single-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nicotinamide mononucleotide (NMN-C) (Experimental): Nicotinamide mononucleotide (NMN-C) at 400 mg/day for 28 days in total
  Interventions: Dietary Supplement: Nicotinamide mononucleotide (NMN-C)

INTERVENTIONS:
Dietary Supplement: Nicotinamide mononucleotide (NMN-C) — Nicotinamide mononucleotide (NMN-C) at 400 mg/day for 28 days in total

SUMMARY:
The purpose of this study is to evaluate the physiological and/or biological actions of nicotinamide mononucleotide (NMN-C) in healthy adults receiving a repeated-dose over the course of 28 days by studying the tolerance and pharmacodynamics of this product.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers should be

* Men between the ages of 30 and 60 years old
* With a BMI between 23 and 30 kg/m2
* With a weight > or = 70kg
* Giving their free informed consent to the study

Exclusion Criteria:

May not be included in the study Volunteers with

* a history of allergy to vitamin B3 (niacin or nicotinamide)
* immunocompromised or suffering from a serious or progressive disease (cardiac, pulmonary, hepatic, renal, hematologic, neoplastic or infectious)
* with abnormal results on the screening bioassay (CBC, Transaminases (AST, ALT, GGT), Bilirubin, Creatinine, CPK, Ionogram, Blood glucose, Hba1c, Lipid profile)
* having donated blood in the month preceding inclusion,
* having consumed more than 2 glasses of alcohol per day,
* being under medication or taking food supplements,
* having reached the maximum compensation threshold for research involving the human being as provided for by the regulations or having participated in another biomedical research project that required blood samples in the previous month,
* involved in another clinical trial or being in the exclusion period of a previous clinical trial.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in NAD+ concentrations in whole blood | Day 0, Day 14 and Day 28

SECONDARY OUTCOMES:
Change from baseline in NMN concentrations in whole blood | Day 0, Day 14 and Day 28
Change from baseline NAD+ metabolite concentrations in plasma | Day 0, Day 14 and Day 28
  MeNAM, NAM, DMG, TMG and Homocystein
Change from baseline NAD+ metabolite concentrations in urine | Day -7, Day 14 and Day 28
  MeNAM and Me-2-PY
Adverse events | Day 14 and Day 28
  Evaluation of adverse events
Evolution of the mitochondrial DNA ratio | Day 0 and Day 28
  mitochondrial DNA ratio will be assessed in the epithelial cells collected by buccal swabs
Evolution of blood glucose levels | Day -7, Day 14 and Day 28
Evolution of blood lipid levels | Day -7, Day 14 and Day 28
  Triglycerides, Total Cholesterol, HDL-Cholesterol, LDL-Cholesterol
Evolution of Transaminases (ASAT, ALAT, GGT) levels in blood | Day -7, Day 14 and Day 28
Evolution of Blood cell count | Day -7, Day 14 and Day 28
Evolution of Bilirubin levels in blood | Day -7, Day 14 and Day 28
Evolution of Creatinine levels in blood | Day -7, Day 14 and Day 28
Creatine phosphokinase (CPK) levels in blood | Day -7, Day 14 and Day 28
Evolution of blood Ionogram | Day -7, Day 14 and Day 28
  Potassium, Chloride, Sodium levels will be assessed in blood
Evolution of Diastolic blood pressure | Day -7 and Day 28
Evolution of Systolic blood pressure | Day -7 and Day 28
Evolution of Heart rate | Day -7 and Day 28
Evolution of weight | Day -7, Day 14 and Day 28
Evolution of body composition | Day -7, Day 14 and Day 28
  Body composition will be assessed by impedancemetry

CONTACTS AND LOCATIONS:
Locations (1):
- Biomed 21, Dijon, France

IPD SHARING:
Plan to Share IPD: No